CLINICAL TRIAL: NCT04326322
Title: Methionine Requirements During Healthy Human Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Rajavel Elango, PhD, Principal Investigator, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: H20-00383
Record Dates: First submitted 2020-03-26; First posted 2020-03-30 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Pregnancy Related
Keywords: nutrition; methionine; sulfur amino acids; stable isotope

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Methionine Intake (Experimental): Oral consumption of eight hourly experimental meals- Includes 4 tracer-free experimental meals containing a mixture of free amino acids, calories from a flavored liquid and protein free cookies and 4- labeled amino acid experimental meals.
  Interventions: Dietary Supplement: Methionine Intake

INTERVENTIONS:
Dietary Supplement: Methionine Intake — Intakes will be randomly chosen from a list of 7 doses of methionine. Each intake will will be repeated approximately 5 times.

SUMMARY:
The current recommendations for dietary amino acid intake in pregnant women are based on calculations from requirements of adult men. The study aims to determine methionine requirements during early (11-20 weeks) and late (31-38 weeks) stages of pregnancy. Methionine, an essential amino acid (building block of body protein), is necessary for protein synthesis and for DNA related cellular functions. A non-invasive, novel method based on different diets, stable isotopes (the safe kind) and simple breath collection will be used. This method has recently been used by our laboratory to study other amino acids during pregnancy.

DETAILED DESCRIPTION:
Pre-study day protocol:

Participants will be asked to meet for a brief (1 hour) pre-study assessment in preparation for the study day. Participants' eligibility will be assessed during this time. Subjects will arrive at the British Columbia Children's Hospital Research Institute's Clinical Research and Evaluation Unit (CREU) having fasted overnight (at least 8 hours since last caloric intake; no morning exercise, and assisted transportation to minimize stress). The consent form will be thoroughly explained, with the subject instructed to stop and ask questions at any point in which they are confused or uncomfortable. If the participants are willing to participate, verbal consent and a signature will be obtained. On this day, participants will fill out a questionnaire, and the following measurements will be taken: height (Harpenden Stadiometer; Holtain Limited, UK) and weight (electric scale; HealthOMeter Professional, Sunbeam Products, Inc.), bioelectrical impedance analysis (BIA; Q4 Bioimpedance Analyzer, RJL Systems, MI), 3 site skinfold (Harpenden Calipers; Baty International, UK), blood glucose (One Touch Ultra, LifeScan, Inc.), and resting energy expenditure (REE; Vmax Encore, Viasys, CA). The REE describes the caloric requirement for vital function in the absence of physical exertion. This value will be used to calculate the total energy content of the experimental diets in order to ensure that the specific caloric needs of each participant will be met. Blood glucose will be assessed for gestational diabetes mellitus (GDM; fasting plasma glucose level of 5.3 mmol/L indicative of GDM). Skinfold and BIA measurements will be collected to determine maternal fat and fat free mass.

Study day protocol:

Healthy pregnant women (20-40 y) who have consented and participated in the pre-study day will be studied at two stages of gestation (n=15/stage) over a range of test methionine intakes (ranging from 0-40mg/kg/day). At the beginning and end of the day a urine dipstick test will be performed. Each study day will be separated by a week and will receive a different, random methionine test intake. On the day of the study, participants will come in fasted at ~8 am for a total of eight hours. They will receive eight hourly meals, which represent 1/12 of their balanced nutritional need for the day. The meals consist of an orange flavoured shake with egg protein composition, balanced with sufficient carbohydrates and lipids. A tracer amino acid (L-[1-13C] phenylalanine) will be provided with the test meals to assess oxidation of the tracer to 13CO2 (13C- carbon dioxide) in breath in response to the test/limiting amino acid (methionine). Open-circuit indirect calorimetry will be performed until 5 steady state data points will be obtained for the measurement of VCO2 (Carbon Dioxide Output; Vmax Encore, Viasys, CA). This technique, called the indicator amino acid oxidation method, is a novel, non-invasive and completely safe approach especially in pregnancy.

Throughout the 8-hour study period biological samples (breath, urine, blood) will be collected and analyzed for 13CO2 content and sulfur amino acid metabolites.

ELIGIBILITY:
Inclusion Criteria:

1. Women who are 20-40 years of age. This includes women of reproductive age who have a low relative risk ratio of maternal or neonatal morbidities.
2. Women pregnant with a singleton pregnancy.
3. Women who are 11-20 or 31-40 weeks pregnant.
4. In apparently good health. Subjects must not have pre-existing health conditions.

Exclusion Criteria:

1. Women who are not pregnant or who are pregnant with more than one fetus.
2. Women who were pregnant in the 6 months before the current pregnancy
3. Women with history of spontaneous abortion (within the last 6 months) or pre-term birth
4. Women who are younger than 20 years of age and older than 40 years of age.
5. Women with a metabolic, neurological, genetic or immune disorder likely to affect nutritional requirements or overall body metabolism.

5. Women who depend on medication that affects normal metabolism. 6. Women experiencing severe nausea, food avoidance or vomiting throughout their pregnancy.

7. Women allergic to eggs or egg protein. 8. Women classified as underweight (<18.5 kg/m2), overweight (25-30 kg/m2) or obese (>30 kg/m2).

9. Women smoking cigarettes, taking illicit drugs, or consuming alcohol regularly during their pregnancy.

10. Women who do not take a prenatal vitamin for the duration of their study period.

11. Women who have lost weight (approximately 1.5kg or more) during their current pregnancy.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 69 (Actual)
Dates: Start 2020-09-14 (Actual); Primary Completion 2023-06-21 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
The rate of oxidation of 13C phenylalanine. | 8 hours
  Urine, breath and a single blood sample will be collected during the study to measure the rate of oxidation of 13C phenylalanine.

CONTACTS AND LOCATIONS:
Overall Officials: Rajavel Elango, PhD, Principal Investigator — University of British Columbia
Locations (1):
- BC Children's Hospital Research Institute, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Scherbinsky K, Rasmussen BF, Li B, Kong D, Ball RO, Pencharz PB, Courtney-Martin G, Elango R. Total sulfur amino acid requirements are higher during late gestation compared with early gestation in healthy Canadian pregnancies in a repeated-measures trial. Am J Clin Nutr. 2024 Oct;120(4):973-983. doi: 10.1016/j.ajcnut.2024.07.034. Epub 2024 Aug 10. PMID 39128498